CLINICAL TRIAL: NCT07367217
Title: Albumin Platelet-Rich Fibrin in Lateral Sinus Floor Augmentation With Simultaneous Implant Placement: A Prospective Two-Year Follow-Up Study
Brief Title: Albumin-PRF in Sinus Lift With Implants: 2-Year Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ammar Radwan, postgraduate student, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R.25.12.93
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sinus Lift Augmentation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lateral sinus lift with bone augmenation (Experimental)
  Interventions: Procedure: lateral sinus lift with using allograft and pericardium membrane
- lateral sinus lift with extended platelet rich fibrin (Experimental)
  Interventions: Procedure: lateral sinus lift with using exteneded platelet rich fibrin

INTERVENTIONS:
Procedure: lateral sinus lift with using allograft and pericardium membrane — sinus floor elevation with placing allograft and collagen membrane
  Arms: lateral sinus lift with bone augmenation
Procedure: lateral sinus lift with using exteneded platelet rich fibrin — sinus floor elevation with placing extended-PRF
  Arms: lateral sinus lift with extended platelet rich fibrin

SUMMARY:
thirty-two implants will be inserted in patients seeking implantation of their lost posterior maxillary teeth (premolar and molars) with limited bone height below the floor of the maxillary sinus, secondary to sinus pneumatization. The patients will be selected from those attending the outpatient clinic of the Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Mansoura University.

ELIGIBILITY:
Inclusion Criteria:

* Patent ostium of maxillary sinus.
* Patient with missing one or more posterior maxillary teeth.
* Residual bone height of 3-6 mm, measured from the crest of alveolar ridge to the floor of the maxillary sinus at the planned implant site.
* A ridge width at the site of implantation of <5mm.
* Platelets of normal range.
* Good oral hygiene.
* Patients in the age frame between 20 years and 60 years old.
* No gender preface in selection of the patients.
* A minimum crown height space of 8 mm.

Exclusion Criteria:

* Active sinusitis, cyst, tumors or root tips at the planned surgical site.
* Patients with systemic diseases that contra-indicate the surgical procedure such as uncontrolled diabetes mellitus, bleeding disorders, serious osseous disorders, and mental disorders.
* Heavy smoking and alcoholism.
* Parafunctional habits such as bruxism and clenching.
* Signs of acute infection or pus discharge.
* Disturbed occlusion.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
1. implant stability | 12 months
  the stability of the implants will be evaluated by RFA with the Osstell Mentor device.
2. Vertical bone height | 24 Months
  vertical bone height will be measured as the distance from the alveolar crest to the new sinus floor at the middle of the implant

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt